CLINICAL TRIAL: NCT02202330
Title: Translating Knowledge for Action Against Stroke - Using 5 Minute Videos for Numeracy and Literacy Challenged Stroke Survivors and Caregivers to Improve Outcomes
Brief Title: Using 5 Minute Videos for Numeracy and Literacy Challenged Stroke Survivors to Improve Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor Neurology,Director Stroke Services, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: URC132001MED
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care, Organized Discharge (Placebo Comparator): Stroke patients are given instructions before discharge regarding diet, need for rehabilitation, possible complications, medication use and information booklets are also handed out. This information is imparted by a multidisciplinary team consisting of a neuro physician, a stroke nurse, a dietitian and a physiotherapist. These are verbal instructions and handouts are written in English. On the day of discharge, or 24 hours prior to discharge, a discharge coordinator details the skills learnt . A detailed written discharge summary is given out detailing all aspects of care, follow-up, medications and test results.
  Interventions: Other: Video Arm
- Video Arm, Standard Discharge (Experimental): Intervention is as follows:
  1. 5 minute videos, on various stroke related topics/ themes delivered in one session before discharge from the hospital (list topics on which videos have to made)
  2. Discussion and questions and answers after viewing video to ensure that core message has been understood and there are no lacunae in understanding the message of video.
  3. Phone card - a memory chip installed in the cell phones of intervention team that ensures that the videos can be replayed at home to refresh memory of some details that may not have been captured in the mandatory viewing sessions.
  Interventions: Other: Video Arm

INTERVENTIONS:
Other: Video Arm — 1. 5 minute videos, on various stroke related topics/ themes delivered in one session before discharge from the hospital (list topics on which videos have to made)
  2. Discussion and questions and answers after viewing video to ensure that core message has been understood and there are no lacunae in understanding the message of video.
  3. Phone card - a memory chip installed in the cell phones of intervention team that ensures that the videos can be replayed at home to refresh memory of some details that may not have been captured in the mandatory viewing sessions.

SUMMARY:
Two thirds of all strokes happen in developing countries like Pakistan. There is a serious lack of health literacy regarding survival after stroke. We hypothesize that our set of 5 minute videos that teach important skills to stroke survivors and their caregivers , that can be replayed in cell phones for extended learning, will increase their adherence to Medications after stroke and improve the control of blood pressure, elevated cholesterol and glucose in the participants getting cell phone based educational videos.

DETAILED DESCRIPTION:
In 80% of patients with stroke, further events may be prevented by altering lifestyle behavioral risk, and increasing adherence to medications to control hypertension, diabetes, lipids. Yet, there exists a huge science to implementation gap to adopt these widely recognized beneficial medicines and lifestyle changes. Those most in need remain unable to actualize the benefits of science, due to lack of knowledge, perceived complexity, literacy challenges, limited time by poorly communicating doctors in crowded clinics and essentially, failure by regional scientists to translate Western science in creative resonant ways that enable wider uptake.

In this randomized double blind translational implementation study, we will study the effectiveness of the implementation tactic of delivering enabling stroke education and risk reduction to literacy and numeracy challenged Pakistani stroke survivors and their caregivers, via short films teaching stroke recognition, healthy habits, medication adherence and self-care. These 5 minute films , using a 'show me not tell me ' approach, will be replayed in tablets, and shown to all stroke patients in the intervention arm. The primary objective of this study is to answer the research question - Does video based education given to stroke patients (with mild to moderate disability) and their caregivers before discharge, and during follow up, improve adherence to therapy and control of three major risk factors (Diabetes, hypertension and dyslipidemia) at twelve months post index stroke?

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women, > 18 years of age
2. Resident of Karachi and planning to live in Karachi to complete long term follow up
3. Able to understand Urdu (language of the videos)
4. Admitted with first ever stroke (ischemic or hemorrhagic)
5. Modified Rankin score <3 ( Mild strokes)
6. Have at least one vascular risk factor that requires medical intervention
7. Consent to participate in the study and follow up, both stroke and caregiver.
8. Have a stable surrogate caregiver at home who is responsible for appointments, follow-ups, overall care, e.g., wife, daughters, daughter- in- law, etc.

Exclusion Criteria:

1. Serious aphasia, visual hemi neglect, short term memory loss in the patient precluding understanding, visualization or retention of the video material, despite overall "a small stroke", this would be a cognitively critical stroke.
2. Serious aphasia, visual hemi neglect, short term memory loss, dementia in the caregiver precluding understanding, visualization or retention of the video material.
3. Iatrogenic stroke, stroke due to non-atherosclerotic vascular disease and rare causes e.g. moya moya, carotid dissections, gunshot to neck, post Coronary Artery Bypass surgery etc.
4. Serious concurrent medical illnesses, like cancer, renal failure, acute liver disease in past 6 months (that precludes use of statins), chronic liver disease, that exclude the use of stroke preventive medications, or require non standardized therapy.
5. Any use of off label, non-guideline medications, due to patient unique comorbid conditions that interfere with medication compliance to antihypertensive, statins, antiplatelet agents and diabetes control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Increase in Adherence and Control of Stroke Risk Factors | 1, 3, 6, 9 and 12 months
  1. Proportion of participants adhering to medications prescribed (Definition of adherence- use of prescribed medications on >5 days a week and measured by the Morisky adherence scale(18).
  2. Proportion of participants achieving control of blood pressure (control is defined as BP<125/85), blood sugar (HbA1c<7) and blood cholesterol (LDL < 100)(19).

SECONDARY OUTCOMES:
Increase in Knowledge and Decrease in Complications | 1, 3, 6, 9 and 12 months
  1. Increase in knowledge of caretakers concerning stroke risk factors, stroke rehabilitation and medications (A knowledge questionnaire will be designed to cover all aspects. This will be administered at 1, 3, 6, 9 and 12 months and improvement in score will be ascertained).
  2. Readmission to hospital with any of the stroke related complications - Urinary Tract infection, pneumonia, Deep vein Thrombosis (This information will be elicited at the follow-up time, based on recall. All subjects will be asked to bring documents related to any hospital admissions in the period following discharge )

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ayeesha K Kamal, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Clinical Trial Unit, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Kamal A, Khoja A, Usmani B, Magsi S, Malani A, Peera Z, Sattar S, Ahmed Akram M, Shahnawaz S, Zulfiqar M, Muqeet A, Zaidi F, Sayani S, Artani A, Azam I, Saleem S. Effect of 5-Minute Movies Shown via a Mobile Phone App on Risk Factors and Mortality After Stroke in a Low- to Middle-Income Country: Randomized Controlled Trial for the Stroke Caregiver Dyad Education Intervention (Movies4Stroke). JMIR Mhealth Uhealth. 2020 Jan 28;8(1):e12113. doi: 10.2196/12113. PMID 32012080
- [Derived] Kamal AK, Khoja A, Usmani B, Muqeet A, Zaidi F, Ahmed M, Shakeel S, Soomro N, Gowani A, Asad N, Ahmed A, Sayani S, Azam I, Saleem S. Translating knowledge for action against stroke--using 5-minute videos for stroke survivors and caregivers to improve post-stroke outcomes: study protocol for a randomized controlled trial (Movies4Stroke). Trials. 2016 Jan 27;17:52. doi: 10.1186/s13063-016-1175-x. PMID 26818913